CLINICAL TRIAL: NCT05751616
Title: Effect of Speed Sintering on Translucency and Microstructure of High Versus Low Translucent Zirconia Veneers: a Randomized Clinical Trial
Brief Title: A Clinical Trial of the Impact of Speed and Conventional Sintering on Ultra-thin, Highly Translucent, Multilayered Zirconia Laminate Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TP_22
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Dental Veneers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional sintering (Active Comparator)
  Interventions: Other: Laminate veneers with conventional sintering
- Speed sintering (Experimental)
  Interventions: Other: Laminate veneers with speed sintering

INTERVENTIONS:
Other: Laminate veneers with speed sintering — Zirconia specimens will be sintered using speed sintering cycle in a conventional furnace according to the manufacturer instructions.
  Arms: Speed sintering
Other: Laminate veneers with conventional sintering — Zirconia specimens will be sintered using conventional sintering cycle in a conventional furnace according to the manufacturer instructions.
  Arms: Conventional sintering

SUMMARY:
A Minimally invasive esthetic restorative approach with the advancement of highly translucent multilayered monolithic zirconia ceramic can provide minimal thickness that affords high strength and esthetics without the need for layering porcelain. The effect of sintering conditions on yttria-partially stabilized zirconia is essential for the long-term success of such restorations.

The study aims to evaluate the clinical performance of speed and conventional sintering on ultra-thin, highly translucent, multilayered zirconia laminate restorations with minimum invasive tooth preparation.

ELIGIBILITY:
Inclusion Criteria:

* patients able to understand and sign the informed consent form.
* physically and psychologically able to undergo conventional restorative procedures.
* Good oral hygiene with no signs of periapical pathology or periodontal disease. (periodontal screening index 0-1).
* Slight malposition.
* Teeth with spacing.
* Teeth with discoloration.
* Patient having natural teeth as opposing dentition

Exclusion Criteria:

* Insufficient surface enamel (60%).
* Abutments with subgingival restorations or root caries.
* Parafunctional habits.
* Lack of opposite occluding dentition in the area intended for restoration.
* mandibular prognathism and maxillary retrognathism

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in clinical performance | Baseline, 3 months, 6 months, 9 months, 12 months
  Patients will be recalled every 3 months for one year follow up. The clinical evaluation and color measurement will be based on the modified California Dental Association (CDA)/Ryge criteria of evaluation as shown
  Examiners will evaluate the zirconia Veneers for the following:
  1. Color match.
  2. Zirconia surface.
  3. Marginal discoloration.
  4. Marginal integrity.
  5. Clinical evaluation of the completed restorations will be performed using a double-blind assessment method

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinics of Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt